CLINICAL TRIAL: NCT00317213
Title: Phase IIB Study of the Efficacy and Safety of LIBERTAL, A Phosphatidic-Acid-Enriched Phospholipid, on Smoking Cessation
Brief Title: Smoking Cessation Assistance With LIBERTAL, A Phospholipid Mixture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Collaborators: Modus Biological Membranes, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIB-05-2001
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Smoking
Keywords: Smoking; Nicotine; Withdrawal; Phospholipids; Cell membrane fluidity; Smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

INTERVENTIONS:
Drug: LIBERTAL- a phospholipid mixture

SUMMARY:
It has been shown in rodent models that chronic substance abuse is associated with a rigidification of cell membrane fluidity due to a change in the membrane cholesterol/phospholipids ratio. Upon substance withdrawal the membrane undergoes reequilibration of this ratio, a process resulting both in an acute and a prolonged severe withdrawal syndrome. MBM has developed a patented,phosphatidic acid-enriched phospholipid platform ("LIBERTAL"), which is supposed to facilitate the membrane fluidity recovery. The company has focused on nicotine withdrawal in smoking cessation,as primary target.

DETAILED DESCRIPTION:
A randomized,double-blind, dose-finding,phase IIB study with Libertal has been performed in 493 volunteer smokers, wishing to quit. They were divided into 5 arms: 4 treatment groups of 0.5, 1.0, 2.0 and 4.0g/day respectively, and one placebo, divided BID. Treatment was administered during one week prior to smoking cessation, then continued during 8 weeks (56 days), followed by another 4 weeks without treatment (up to day 84). The primary endpoint was complete smoking cessation during at least 28 consecutive days. There were 6 on-site visits and 4 telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Smokers of at least 1 year duration
* Smoking at least 10 cigarettes/day
* Having failed at least one previous smoking cessation effort.
* Without a major cardio-vascular or metabolic disease or condition.

Exclusion Criteria:

* An uncontrolled major cardiovascular, metabolic, or other condition condition.
* Need for surgery during the period of participation in the trial.
* Any treatment for smoking cessation during the 2 months preceding enrollment in the present trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-02; Study Completion 2002-07

PRIMARY OUTCOMES:
Quit Smoking Rates - QSR% as confirmed by CO measurement in exhaled air.
Safety as expressed by adverse-event reporting, clinical, hematological and biochemical parameters.

SECONDARY OUTCOMES:
Immunomodulatory potential of Libertal, as expressed by cytokine measurements in frozen cultured PBMC supernatants

CONTACTS AND LOCATIONS:
Overall Officials: Zeev T. Handzel, M.D., Principal Investigator — Kaplan Medical Center; Avner Shenfeld, Ph.D,, Study Director — Modus Biological Membranes
Locations (1):
- Arazi Clinic and Modus Clinic, Tel-Aviv and Rehovot, Israel